CLINICAL TRIAL: NCT03914755
Title: A Phase 1, Open Label, Safety, Tolerability, and Pharmacokinetic Study of Tucatinib (ONT-380) in Healthy Japanese and Caucasian Subjects
Brief Title: A Safety, Tolerability, and Pharmacokinetic Study of Tucatinib in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNTUC-015
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 50 mg twice daily on Days 1-13 and once daily on Day 14
  Interventions: Drug: Tucatinib
- Cohort 2 (Experimental): 150 mg twice daily on Days 1-13 and once daily on Day 14
  Interventions: Drug: Tucatinib
- Cohort 3 (Experimental): 300 mg twice daily on Days 1-13 and once daily on Day 14
  Interventions: Drug: Tucatinib

INTERVENTIONS:
Drug: Tucatinib — Administered via oral tablet

SUMMARY:
This study is being done to compare the pharmacokinetics (PK) and safety/tolerability of tucatinib in healthy Japanese and Caucasian participants.

Three cohorts of healthy Japanese and Caucasian men and women will be admitted to the Clinical Research Unit (CRU) and receive multiple oral doses of tucatinib over 14 days with and without food.

Subjects will be in the study for up to 45 days, including the screening period.

Due to practical considerations, each cohort will be dosed sequentially (this is not a dose escalation study).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 32 kg/m^2 and a total body weight between 50 and 100 kg
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiograms, vital signs measurements, or clinical laboratory evaluations
* Female subjects participating in the study will be of non-childbearing potential. Male subjects will be surgically sterile for at least 90 days or will agree to use contraception during the study and for 90 days after last dose of study drug.
* Japanese subjects:

  1. Must have been born in Japan
  2. Must have 2 biological Japanese parents and 4 biological Japanese grandparents as confirmed by interview
  3. Must have spent less than 10 years outside of Japan, and has no significant changes in lifestyle, including diet, since leaving Japan

Exclusion Criteria:

* Significant history of metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* Current condition possibly affecting drug absorption
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection that would potentially alter absorption or excretion of orally administered drugs
* History of alcoholism or drug/chemical abuse within 2 years of check-in
* History of regular alcohol consumption exceeding 7 drinks/week for female subjects or 14 drinks/week for male subjects
* Positive hepatitis panel and/or positive human immunodeficiency (HIV) test
* Liver function tests, serum creatinine, hemoglobin, or hematocrit values outside of the normal reference range
* Single 12-lead ECG demonstrating QTcF>450 msec for males or >470 msec for females
* Participation in a clinical study involving administration of an investigational drug in the past 30 days from last dose or 5 half-lives (whichever is longer)
* Use of any products known to alter drug absorption, metabolism or elimination processes, including St. John's wort and known strong inhibitors or inducers of CYP3A4 or CYP2C8, within 30 days
* Use of or intention to use any prescription or nonprescription products, including vitamins, minerals and herbal preparations within 14 days
* Use of tobacco- or nicotine-containing products within 3 months
* Receipt of blood products within 2 months
* Donation of blood from 56 days before the Screening Visit, plasma from 2 weeks before the Screening Visit or platelets from 6 weeks before the Screening Visit
* Poor peripheral venous access
* Have previously completed or withdrawn from this study or any other study investigating tucatinib and have previously received the study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-08-04 (Actual); Study Completion 2019-08-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of tucatinib | 14 days
Cmax of ONT-993 | 14 days
Time of the maximum observed concentration (tmax) of tucatinib | 14 days
Tmax of ONT-993 | 14 days
AUC from time 0 to the time of last quantifiable concentration (AUClast) of tucatinib | 14 days
AUClast of ONT-993 | 14 days
AUC from time 0 to 12 hours postdose (AUC0-12hr) of tucatinib | 14 days
AUC0-12hr of ONT-993 | 14 days
AUC from time 0 extrapolated to infinity (AUC0-inf) of tucatinib | 1 day
AUC from time 0 extrapolated to infinity (AUC0-inf) of ONT-993 | 1 day
Percentage of AUC0-inf due to extrapolation (%AUCextrap) of tucatinib | 1 day
%AUCextrap of ONT-993 | 1 day
Apparent total clearance (CL/F) of tucatinib | 14 days
Apparent volume of distribution during the terminal phase (Vz/F) of tucatinib | 14 days
Metabolite-to-parent molar ratio based on AUC (MRAUC) of ONT-993 | 14 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Woolery, PharmD, BCOP, Study Director — Seagen Inc.
Locations (1):
- PAREXEL International, Early Phase Clinical Unit - Los Angeles, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang D, Taylor A, Zhao JJ, Endres CJ, Topletz-Erickson A. Population Pharmacokinetic Analysis of Tucatinib in Healthy Participants and Patients with Breast Cancer or Colorectal Cancer. Clin Pharmacokinet. 2024 Oct;63(10):1477-1487. doi: 10.1007/s40262-024-01412-0. Epub 2024 Oct 5. PMID 39368039